CLINICAL TRIAL: NCT06065254
Title: Efficacy of Gingival Grafts During the Implantation Process in the Increasing of Peri-implant Keratinized Tissue Width and Soft Tissues Thickness
Brief Title: Efficacy of Gingival Grafts During the Implantation Process on the Peri-implant Mucosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-Perio-01-2023
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Dental Implants; Transplants
Keywords: Keratinized Mucosa; Connective Tissue Graft; Free Gingival Graft

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Free gingival graft (Experimental): Free gingival graft will be applied and and followed for 3 months
  Interventions: Other: Efficacy of free gingival grafts during in the increasing of peri-implant keratinized tissue width and soft tissues thickness
- Connective tissue graft (Experimental): Connective tissue graft will be applied and and followed for 3 months
  Interventions: Other: Efficacy of connective tissue grafts during in the increasing of peri-implant keratinized tissue width and soft tissues thickness
- No grafts will be applied. (Other): No grafts of any types will be applied.
  Interventions: Other: No types of grafts will be made to improve the quality of the peri-implant mucosa

INTERVENTIONS:
Other: Efficacy of free gingival grafts during in the increasing of peri-implant keratinized tissue width and soft tissues thickness — Two vertical incisions will be made in the previously elevated flap against the placed implant , where these two incisions will be 10 mm apart from each other, and the free graft to will be placed in this distance (10 x 10 mm). The graft will be obtained from the donor site (the hard palate), and will be thinned to obtain a regular graft with the required thickness. After that, the graft will be moved to its correct place accurately, while avoiding leaving a distance between the graft and the tissue underneath, and the graft will be sutured well to ensure its stability and correct placement.
  Arms: Free gingival graft
Other: Efficacy of connective tissue grafts during in the increasing of peri-implant keratinized tissue width and soft tissues thickness — Vertical incisions will not be made in the previously elevated flap against the placed implant, where there is no need to suture the flap apically of the grafting place because the graft will be covered with it after fixing it in place. The area will be washed with the serum to remove the clot before fixing the graft.The graft will be obtained from the donor site according to the previously mentioned method. Then the epithelium will be removed to leave the connective tissue underneath, and then the graft will be moved to its place (buccally dental implant site) and the flap will be sutured over it.
  Arms: Connective tissue graft
Other: No types of grafts will be made to improve the quality of the peri-implant mucosa — The simple suturing of the two surgical incisions will be done after the completion of the dental implant process, with no procedure will be made to improve the quality of the peri-implant mucosa.
  Arms: No grafts will be applied.

SUMMARY:
This study aims to compare the changes in the peri-implant mucosa during the application of two soft tissue grafting methods, which are free gingival graft (FGG) and connective tissue graft (CTG) taken from the palatine in terms of the width of the keratinized mucosa and the thickness of the peri-implant soft tissues.

DETAILED DESCRIPTION:
The presence of adequate width of the keratinized gingiva may be necessary in some special cases such as the presence of fixed prostheses on the teeth with sublingual margins or peri implants. There is an association between insufficiency of the keratinized tissues peri implants with greater plaque accumulation, signs of inflammation, soft tissue recession, and loss of attachment. The sample will consist of 33 dental implant sites and divide randomly into three groups: Group I (Experiential, n=11): FGG; Group II: (Experiential, n=11): CTG; and Group III: (Control, n=11): No procedure will be done to improve the quality of the peri-implant tissues. The width of the keratinized gingiva will be measured preoperative with a UNC-15 and the thickness of the peri-implant soft tissues will be measured clinically by direct transgingival propping method. These measurements will be repeated after 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. patients who have lost posterior teeth (premolars or molars).
2. A decrease in the amount of keratinized gingiva (less than 2 mm from the alveolar process to the mucogingival junction).
3. good oral health (plaque index ≤1).

Exclusion Criteria:

1. heavy smokers (more than 10 cigarettes per day)
2. uncontrolled diabetes or other systemic diseases.

Ages: 21 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
The width of the keratinized gingiva | after 1 month and 3 months
  The width of the keratinized gingiva will be measured using a UNC-15 probe from the middle of the alveolar process at the site studied to the mucogingival junction, which was determined by the rollover technique.
The thickness of the peri-implant soft tissues | after 1 month and 3 months
  The thickness of the peri-implant soft tissues will be measured clinically by the direct transgingival propping method.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Alshouaa, MSc, Principal Investigator — MSc student in Periodontology Departement, University of Damascus; Mohammed Alsabbagh, Study Chair — Professor of Periodontology, Department of Periodontology, University of Damascus
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Angelis P, De Angelis S, Passarelli PC, Liguori MG, Pompa G, Papi P, Manicone PF, D'Addona A. Clinical comparison of a xenogeneic collagen matrix versus subepithelial autogenous connective tissue graft for augmentation of soft tissue around implants. Int J Oral Maxillofac Surg. 2021 Jul;50(7):956-963. doi: 10.1016/j.ijom.2020.11.014. Epub 2020 Dec 2. PMID 33279377
- [Background] Schmitt CM, Bruckbauer P, Schlegel KA, Buchbender M, Adler W, Matta RE. Volumetric soft tissue alterations in the early healing phase after peri- implant soft tissue contour augmentation with a porcine collagen matrix versus the autologous connective tissue graft: A controlled clinical trial. J Clin Periodontol. 2021 Jan;48(1):145-162. doi: 10.1111/jcpe.13387. Epub 2020 Nov 12. PMID 33047372
- [Background] Raoofi S, Asadinejad SM, Khorshidi H. Evaluation of Color and Width of Attached Gingiva Gain in Two Surgical Techniques: Free Gingival Graft and Connective Tissue Graft Covered By Thin Mucosal Flap, a Clinical Trial. J Dent (Shiraz). 2019 Dec;20(4):224-231. doi: 10.30476/DENTJODS.2019.44916. PMID 31875168
- [Background] Happe A, Stimmelmayr M, Schlee M, Rothamel D. Surgical management of peri-implant soft tissue color mismatch caused by shine-through effects of restorative materials: one-year follow-up. Int J Periodontics Restorative Dent. 2013 Jan-Feb;33(1):81-8. doi: 10.11607/prd.1344. PMID 23342350
- [Background] Thoma DS, Buranawat B, Hammerle CH, Held U, Jung RE. Efficacy of soft tissue augmentation around dental implants and in partially edentulous areas: a systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S77-91. doi: 10.1111/jcpe.12220. PMID 24641003